CLINICAL TRIAL: NCT02577939
Title: Evaluation of Cardiorespiratory Performance After Interval Exercise Training (IET) Prior to Hematopoietic Cell Transplantation
Brief Title: Evaluation of Cardiorespiratory Performance After Interval Exercise Training Prior to Hematopoietic Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1311
Record Dates: First submitted 2015-02-20; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Stem Cell Transplantation, Hematopoietic
MeSH Terms: interventions — Exercise; Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interval Exercise Training (IET) (Experimental): This is a single arm study. All patients receive the intervention of 6 weeks of pre-transplant IET, pre- and post-tests, and data collection via FitBit accelerometer and weekly surveys.
  Interventions: Behavioral: Interval Exercise Training (IET)

INTERVENTIONS:
Behavioral: Interval Exercise Training (IET) — This is a single arm study. All patients receive the intervention of 6 weeks of pre-transplant IET, pre- and post-tests, and data collection via FitBit accelerometer and weekly surveys.
  Other Names: Aerobic Training; Aerobic Exercise; Endurance Training

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of a pre-transplant, interval exercise training (IET) intervention, in increasing peak oxygen uptake (VO2peak) scores on cycle ergometry. This study will have a lead-in phase to ensure that IET is feasible in this population. Secondary objectives include documenting the safety of IET in this population, evaluating the correlation of VO2peak with other methods of measuring pre-transplant cardiorespiratory performance, comparing the 6 minute walk distance (6MWD) pre and post IET, and establishing the feasibility of the 6MWD when performed unsupervised by a health care professional.

Eligible patients include 40 evaluable autologous (n=20) and allogeneic (n=20; 10 full intensity and 10 reduced intensity) transplant patients deemed appropriate for exercise intervention by their treating physician. The investigators will enroll no more than 50 patients onto this trial. Results of this study will inform a randomized, multi-site study of a pre-transplant exercise intervention.

DETAILED DESCRIPTION:
The primary purpose of the study is to determine the ability of a pre-transplant exercise intervention to improve cardiorespiratory performance (measured by VO2peak). If the safety of this approach is documented, and its efficacy demonstrated, a foundation will be laid for a larger, randomized, multi-center study to formally determine the benefit of the pre-transplant exercise intervention.

We plan to analyze the effect of IET on VO2peak in the auto and allo groups separately given their different course of treatment and outcomes. Study subjects will be recruited after they and their transplant teams have decided that they will undergo HCT. Following recruitment, patients will undergo baseline fitness assessments and then receive an individualized IET prescription for a duration of 6 weeks prior to stem cell mobilization (auto) or prior to hospitalization for conditioning (allo). For the first two weeks, subjects will undergo three times weekly 3 minute interval training during walking at 60-70% MHR. This will be followed by three times weekly aerobic interval training for 5 three-minute bouts at 65-85% maximum heart rate per session for 4 weeks.

All patients will also be provided with a FitBit accelerometer. Prior to transplant, patients will undergo follow-up fitness assessments. All patients will undergo activity tracking by accelerometry (FitBit) and admission/weekly symptom/HRQOL tracking by electronic survey throughout the post-transplant hospitalization. Also during hospitalization, all patients will perform weekly clinician supervised 6MWD testing while inpatient. One of the weekly tests during hospitalization will include patient self-administered (clinician observed) 6MWD, along with the clinician supervised 6MWD. Unsupervised patient performed 6MWD will be considered feasible if all patients who perform 6MWD can do so safely, and if for 80% of patients, the patient-performed 6MWD values are within 10% of the corresponding clinician supervised 6MWD results. If feasibility is met, we will ask patients to perform the 6MWD weekly for 4 weeks post discharge and record their distance.

ELIGIBILITY:
Inclusion Criteria:

* Not currently participating in IET training
* Willing and able to provide signed, informed consent
* Planned autologous or allogeneic stem cell transplant with schedule that accommodates a 6 week exercise intervention
* Willing to participate in an IET program that will last 6 weeks.
* Subject must complete at least one interval exercise session during the 6 weeks in order to be eligible for analysis.
* Planning to undergo transplant but continuing to receive cycles of chemotherapy on a previously started regimen while awaiting transplant

Exclusion Criteria:

* Dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent
* Received erythropoiesis-stimulating proteins (ESPs) within 4 weeks prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Of those patients with heart rate data, number and percent of patients able to achieve 65-85% heart rate during one or more exercise sessions. Unit of measurement: number of patients and percent of patients with evaluable heart rate data. | During the 6 weeks of IET pre-transplant
  Establish the feasibility of IET in patients prior to autologous or allogeneic transplantation. Feasibility is defined as 5 of the first 10 evaluable patients being able to achieve 65-85% heart rate during one or more exercise sessions throughout the duration of the interval exercise training.

SECONDARY OUTCOMES:
Number of adverse events as reported by patients and determined by study investigators. Unit of measurement: cumulative number of adverse events. | During the 6 weeks of IET pre-transplant
  Documentations of any IET related complications during the 6 week training program
Change in 6 minute walk distance based on pre- and post- intervention 6 minute walk distance testing. Unit of measurement: meters. | Pre- and Post- Assessment for 6 weeks of IET
  Evaluate cardiorespiratory performance as measured via 6MWD pre and post IET
Change in VO2peak based on pre- and post- intervention VO2peak measurement from cardiopulmonary exercise testing. Unit of measurement: ml/kg*min. | Pre- and Post- Assessment for 6 weeks of IET
  Evaluate cardiorespiratory performance as measured via VO2peak pre and post IET

CONTACTS AND LOCATIONS:
Overall Officials: William A Wood, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States